CLINICAL TRIAL: NCT03842826
Title: Inter-examiner Reproducibility of Clinical Examination Tests for Athletes with Longstanding Groin Pain
Status: Completed | Type: Observational
Sponsor: Aspetar (Other)
Responsible Party: Principal Investigator, Andreas Serner, Principal Investigator, Aspetar
Other Study IDs: Aspetar_GPCA001
Record Dates: First submitted 2019-02-14; First posted 2019-02-15 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Groin Injury; Adductor Strains; Iliopsoas Syndrome
Keywords: Clinical examination; Groin; Reproducibility
MeSH Terms: interventions — Palpation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Athlete: Male athletes performing sports ≥ 1x/week Age: 18-40 years
  Interventions: Diagnostic Test: Palpation, resistance and stretch tests

INTERVENTIONS:
Diagnostic Test: Palpation, resistance and stretch tests — Palpation, resistance and stretch tests performed by 2 blinded examiners.

SUMMARY:
This study will investigate the reproducibility of clinical palpation, resistance and stretching tests which are currently being used for the diagnosis of longstanding groin pain in male athletes.

DETAILED DESCRIPTION:
The "Doha agreement meeting on terminology and definitions" aimed to simplify the heterogeneous taxonomy of groin injuries by creating a straightforward classification system based on patient history and clinical examination. Following this classification system, groin pain can be divided into four defined clinical entities (adductor-, inguinal-, iliopsoas- and/or pubic-related groin pain), hip related groin pain, and/or other causes for groin pain.

In the Doha classification, pain on palpation, resistance and/or stretching are the key clinical findings for categorizing in the four clinical entities. However, this classification does not describe how these clinical tests should be performed and if these tests are reproducible.

The primary aim of this study is to evaluate the inter-examiner reproducibility of clinical palpation, resistance and stretch tests for longstanding groin pain in athletes. The secondary aim is to identify the proportion of positive clinical tests for each clinical entity diagnosis.

Two blinded examiners (a physiotherapist and a general surgeon, both specialized in groin injuries with >10 years experience) will assess each athlete with longstanding groin pain following a standardized examination protocol. Prior to clinical examination, participants will be requested to complete a standardized form for patient/injury characteristics and injury history, the Copenhagen Hip and Groin Outcome Score (HAGOS) and the Oslo Sports Trauma Research Center (OSTRC) overuse injury questionnaire. The HAGOS is a patient-reported outcome measure, which quantifies a patient's current subjective perception of their hip and groin pain within the last week on six subscales, each with a score between 0 and 100.The OSTRC overuse injury questionnaire has a focus on groin problems within the last week.

The standardized clinical examination protocol consists of palpation, resistance and stretch-tests and are used to categorize athletes into defined clinical entities. A score on the Numeric Pain Rating Scale (0-10) will be asked to the patient for each test, where pain during the test has to correspond to the injury pain. Each score from 1-10 will be considered as positive for analysis. If the pain is just from palpation and not related to the injury, the test will be considered negative.

Inter-examiner reliability will be analysed using Cohen's Kappa statistic (κ), including 95% confidence intervals for dichotomous variables. Linear weighted κ will be calculated for ordinal variables. Additionally, the absolute positive agreement and negative agreement between the two examiners and bias index will be calculated. The mean prevalence of each positive clinical tests of both clinicians will be reported for each entity diagnosis. Furthermore, agreement analysis for the palpation tests of the four defined clinical entities of groin pain will also be grouped: adductor-, iliopsoas-, inguinal- (with and without invagination) and pubic palpation.

For the 3 main defined clinical entities (adductor-, inguinal- and iliopsoas-related groin pain), a prevalence is expected between 30-60% in our research population. Assuming that approximately 4 out of every 5 tests (80%) targeting each entity will be positive, we expect a prevalence of positive tests of approximately 24-48% in the whole sample. With an expected Kappa of at least 0.8, with a 95% confidence interval lower limit of 0.4, using a 2-tailed test and assuming no bias between examiners, at least 60 affected sides will be needed for this study. A lower prevalence of positive tests for pubic-related groin pain and subsequent less robust results for clinical tests of this entity will be accepted. No dropout is expected due to the cross-sectional character of the study. We will continue inclusion until we have 60 full data sets.

ELIGIBILITY:
Inclusion Criteria:

* Male athlete (performing sports ≥ 1x/week) with sports-related groin pain ≥ 4 weeks
* Age: 18 - 40 years

Exclusion Criteria:

* Prior assessment/treatment of one of the two examiners for the same complaint (<6 months)
* Prior surgery in the hip- and groin area
* Clinical signs of prostatitis or urinary tract infections
* More than 7 days between the two examiners assessment

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Male athletes with sports-related groin pain ≥ 4 weeks
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Cohen's Kappa statistic (κ) | February 2019 - December 2020
  Inter-examiner reliability

SECONDARY OUTCOMES:
Raw agreement | February 2019 - December 2020
  Absolute positive agreement and negative agreement

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Tol, MD / PhD, Study Director — Aspetar Orthopaedic and Sports Medicine Hospital / Academic Medical Center Amsterdam
Locations (1):
- Aspetar Orthopaedic and Sports Medicine Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided
There is currently no plan of sharing individual participant data; however, upon reasonable request, anonymized data can be made available for interested parties.

REFERENCES:
- [Background] Weir A, Brukner P, Delahunt E, Ekstrand J, Griffin D, Khan KM, Lovell G, Meyers WC, Muschaweck U, Orchard J, Paajanen H, Philippon M, Reboul G, Robinson P, Schache AG, Schilders E, Serner A, Silvers H, Thorborg K, Tyler T, Verrall G, de Vos RJ, Vuckovic Z, Holmich P. Doha agreement meeting on terminology and definitions in groin pain in athletes. Br J Sports Med. 2015 Jun;49(12):768-74. doi: 10.1136/bjsports-2015-094869. PMID 26031643
- [Background] Kottner J, Audige L, Brorson S, Donner A, Gajewski BJ, Hrobjartsson A, Roberts C, Shoukri M, Streiner DL. Guidelines for Reporting Reliability and Agreement Studies (GRRAS) were proposed. Int J Nurs Stud. 2011 Jun;48(6):661-71. doi: 10.1016/j.ijnurstu.2011.01.016. Epub 2011 Apr 23. PMID 21514934
- [Background] Thorborg K, Holmich P, Christensen R, Petersen J, Roos EM. The Copenhagen Hip and Groin Outcome Score (HAGOS): development and validation according to the COSMIN checklist. Br J Sports Med. 2011 May;45(6):478-91. doi: 10.1136/bjsm.2010.080937. PMID 21478502
- [Background] Holmich P, Holmich LR, Bjerg AM. Clinical examination of athletes with groin pain: an intraobserver and interobserver reliability study. Br J Sports Med. 2004 Aug;38(4):446-51. doi: 10.1136/bjsm.2003.004754. PMID 15273182
- [Background] Clarsen B, Myklebust G, Bahr R. Development and validation of a new method for the registration of overuse injuries in sports injury epidemiology: the Oslo Sports Trauma Research Centre (OSTRC) overuse injury questionnaire. Br J Sports Med. 2013 May;47(8):495-502. doi: 10.1136/bjsports-2012-091524. Epub 2012 Oct 4. PMID 23038786
- [Background] Delahunt E, Thorborg K, Khan KM, Robinson P, Holmich P, Weir A. Minimum reporting standards for clinical research on groin pain in athletes. Br J Sports Med. 2015 Jun;49(12):775-81. doi: 10.1136/bjsports-2015-094839. PMID 26031644
- [Background] Thorborg K, Reiman MP, Weir A, Kemp JL, Serner A, Mosler AB, HOlmich P. Clinical Examination, Diagnostic Imaging, and Testing of Athletes With Groin Pain: An Evidence-Based Approach to Effective Management. J Orthop Sports Phys Ther. 2018 Apr;48(4):239-249. doi: 10.2519/jospt.2018.7850. Epub 2018 Mar 6. PMID 29510653
- [Background] Landis JR, Koch GG. The measurement of observer agreement for categorical data. Biometrics. 1977 Mar;33(1):159-74. PMID 843571
- [Background] Taylor R, Vuckovic Z, Mosler A, Agricola R, Otten R, Jacobsen P, Holmich P, Weir A. Multidisciplinary Assessment of 100 Athletes With Groin Pain Using the Doha Agreement: High Prevalence of Adductor-Related Groin Pain in Conjunction With Multiple Causes. Clin J Sport Med. 2018 Jul;28(4):364-369. doi: 10.1097/JSM.0000000000000469. PMID 28654441
- [Derived] Heijboer WMP, Vuckovic Z, Weir A, Tol JL, Holmich P, Serner A. Clinical examination for athletes with inguinal-related groin pain: interexaminer reliability and prevalence of positive tests. BMJ Open Sport Exerc Med. 2023 Jan 11;9(1):e001498. doi: 10.1136/bmjsem-2022-001498. eCollection 2023. PMID 36643406